CLINICAL TRIAL: NCT07084922
Title: Association Between Plantar Pressure Distribution and Postural Balance Parameters in Individuals With Diabetic Foot
Brief Title: An Analysis of Plantar Pressure Distribution and Postural Balance Parameters in Individuals With Diabetic Foot Diagnosis
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Yağmur UYSAL, Lecturer, Medipol University
Other Study IDs: MedipolU-OPZ-YU-02
Record Dates: First submitted 2025-07-02; First posted 2025-07-25 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Diabetes and Risk of Diabetic Foot Ulcer; Diabetes Mellitus; Postural Control; Plantar Pressure Distrubution
Keywords: Postural Control; Diabetic Foot; Plantar Pressure; Plantar Loading
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot | interventions — Postural Balance; Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No interventions. This is an observational study where participants undergo assessments of plantar pressure and postural balance without any treatment or intervention. — No interventions. This is an observational study where participants undergo assessments of plantar pressure and postural balance without any treatment or intervention.

SUMMARY:
This study aims to investigate the relationship between plantar pressure distribution and postural balance in individuals diagnosed with diabetic foot. Diabetic foot is a common and serious complication of diabetes that increases the risk of foot ulcers and falls. Due to nerve damage and changes in walking biomechanics, individuals with diabetic foot may experience abnormal pressure on the soles of their feet and poor balance.

The study includes 32 participants aged 40-65 years who have been clinically diagnosed with diabetic foot (Stage 0 or 1 according to the Meggitt-Wagner classification). Participants undergo plantar pressure assessment using a pedobarographic system and balance testing using a Wii Balance Board system under different standing conditions (eyes open/closed, single/double leg stance). The study aims to identify high-risk plantar regions and impaired balance patterns to guide early interventions, reduce ulcer risk, and prevent falls.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 40 and 65 years
* Diagnosed with diabetic foot at Stage 0 or Stage 1 according to the Meggitt-Wagner classification
* No history of foot or ankle surgery
* Able to walk independently without assistive devices
* Clinically assessed as at risk for diabetic foot

Exclusion Criteria:

* History of amputation in the foot or ankle
* Previous foot or ankle surgery
* Use of medications affecting balance or gait
* Presence of any neurological or musculoskeletal disorder unrelated to diabetic foot that affects mobility or balance

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diagnosed with diabetic foot
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2025-06-28 (Actual); Primary Completion 2025-08-21 (Actual); Study Completion 2025-08-21 (Actual)

PRIMARY OUTCOMES:
Postural balance assessment | first day of the study
  Postural balance assessment in the study will be performed with 'Becure Balance System (Becure Global GmbH)'. Individuals will be evaluated for balance on the device with eyes open-closed, single foot-double foot.
Pedobarographic analysis | first day of the study
  Pedobarographic analysis and evaluation of postural balance are widely used by clinicians and researchers to examine the foot structure and to determine the loading patterns of the foot. The data are obtained with electronic sensors placed on the platform where the gait takes place. The sensors are directly connected to the platforms and the computer system programmed to perform foot analysis. With the pedobarography device, pressure distribution data in the foot are obtained in static condition. Foot plantar pressure analysis will be performed using the EsCoSCAN® static pedobarographic assessment device. During the analysis, the individual will be made to stand without moving while looking straight ahead in the standing position for static analysis.
Demographic Information Form | first day of study
  The patient's demographic information, including height, weight, age, and diabetes type (Type 1 or Type 2), will be recorded using this form. Body Mass Index (BMI) will be calculated based on the recorded height and weight data (BMI = weight [kg] / height² [m²]

CONTACTS AND LOCATIONS:
Overall Officials: yağmur uysal, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
not sure